CLINICAL TRIAL: NCT05556733
Title: Faecal Microbiota Transplantation for Post-acute COVID-19 Syndrome: a Pilot Open-label Study
Brief Title: FMT for Post-acute COVID-19 Syndrome
Acronym: FMT-PACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor Siew Chien NG, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-PACS
Record Dates: First submitted 2022-08-18; First posted 2022-09-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Post-Acute COVID19 Syndrome; COVID-19
Keywords: Faecal Microbiota Transplantation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The intervention group will receive FMT while the control group will not receive FMT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faecal Microbiota Transplantation (Experimental): Subjects will receive Faecal Microbiota Transplantation
  Interventions: Procedure: Faecal Microbiota Transplantation
- Control (No Intervention): The control subjects will not receive FMT

INTERVENTIONS:
Procedure: Faecal Microbiota Transplantation — FMT at baseline, week 2, week 4, week 8
  Arms: Faecal Microbiota Transplantation

SUMMARY:
In recovered COVID-19 patients, emerging global data have reported the presence of long COVID, that is, at least one symptom that an alternative diagnosis cannot explain has been persistent for four or more weeks after the initial infection. We demonstrated previously that almost 80% of recovered COVID-19 patients in Hong Kong suffer from Long COVID for more than 6 months, affecting multiple body systems.

In a recent study, the five most common Long COVID symptoms were fatigue, memory problem, difficulty sleeping, anxiety and hair loss. One promising hypothesis is the involvement of the gut microbiota, a collection of the trillions of gut microorganisms that play important immunomodulatory roles against infections.

Faecal microbiota transplantation (FMT), which is the infusion of processed faeces from healthy donors to the gut of affected subjects, has shown impressive therapeutic effects for recurrent Clostridioides difficile infection and other emerging indications. Gut microorganisms together with the metabolites in the donated faeces could potentially modulate the gut microbiota of the recipient and treat the dysbiosis associated with pathological health conditions. To date, no study has yet to assess the therapeutic effects of FMT in post-COVID-19 neuropsychiatric conditions.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is the disease caused by a novel coronavirus SARS- CoV-2. In recovered COVID-19 patients, emerging global data have reported the presence of Long COVID, a condition where at least one symptom that cannot be explained by alternative diagnosis has been persistent for four or more weeks after the initial infection. We demonstrated previously that almost 80% of recovered COVID-19 patients in Hong Kong suffer from Long COVID for more than 6 months, affecting multiple body systems.

In a recent study, the five most common Long COVID symptoms were fatigue, memory problem, difficulty sleeping, anxiety and hair loss. Current treatment for Long COVID only involves symptomatic care, as the exact mechanisms underlying the pathogenesis are still largely unknown. One promising hypothesis is the involvement of the gut microbiota, a collection of the trillions of gut microorganisms that play important immunomodulatory roles against infections. Our recently published findings have shown that patients with Long COVID had a less diverse gut microbiota with significantly fewer health-associated commensal bacteria than those without Long COVID. Previous studies have also proved the association between the gut microbiota and insomnia, circadian disturbance and affective disorders. Thus, gut microbiota modulation could be a novel therapeutic strategy for these neuropsychiatric conditions.

Faecal microbiota transplantation (FMT), which is the infusion of faeces from healthy donors to the gut of affected subjects, has shown impressive therapeutic effects for various diseases. To date, no study has yet to assess the therapeutic effects of FMT in post-COVID-19 neuropsychiatric conditions. In this pilot open-label study, we aim to explore the efficacy of FMT in improving neuropsychiatric symptoms including but not limited to insomnia severity, sleep quality, anxiety and fatigue in recovered COVID-19 patients. FMT will be administrated via Oesophago-gastro-duodenoscopy (OGD) and Flexible Sigmoidoscopy (FS). Two arms will be recruited in a 1:1 ratio. The intervention group will receive FMT while the control group will not receive FMT. Both groups will have the same assessments. Subjects will receive FMT via OGD at week 0, week 2, week 4 and week 8, and via FS at week 0. Final follow-up will be scheduled at weeks 8 and 12 for clinical assessment. To assess the efficacy of FMT in improving neuropsychiatric symptoms, subjects will have to fill in study questionnaires at baseline, week 8 and week 12. Subjects will also be asked to fill in a sleep diary daily until week 12.

ELIGIBILITY:
Both the interventional group and control group will meet the criteria below and the control group will be age- and sex-matched subjects with the interventional group.

Inclusion Criteria:

* Individuals aged 18 and above
* Subjects who were recovered cases of COVID-19 confirmed by RT-PCR or rapid antigen test (RAT)
* Subjects who had insomnia symptoms of post-acute COVID-19 syndrome at screening visit

Exclusion Criteria:

* Confirmed current active malignancy
* Had abdominal surgery
* Known history of severe organ failure (including decompensated cirrhosis), renal failure on dialysis, suffering from human immunodeficiency virus infection;
* Known pregnancy
* Mental retardation or inability to provide informed consent
* Contraindications to upper GI endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in insomnia severity | 12 weeks
  Severity of insomnia will be measured by a 7-item Insomnia Severity Index (ISI). ISI is a self-report questionnaire used to evaluate the nature, severity and impact of insomnia. Total score ranges from 0 to 28. Higher score indicates more severe insomnia.

SECONDARY OUTCOMES:
Change in sleep quality | 12 weeks
  Quality of sleep will be measured by a 19-item Pittsburgh Sleep Quality Index (PSQI). PSQI is a self-report questionnaire used to evaluate sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Total score ranges from 0 to 21. Lower score indicates healthier sleep quality.
Change in anxiety symptoms | 12 weeks
  Anxiety symptoms will be assessed by a 7-item Generalised Anxiety Disorder-7 scale (GAD-7). GAD-7 is a widely used diagnostic self-report scale for the screening, diagnosis and severity assessment of anxiety disorder. Total score ranges from 0 to 21. Higher score indicates more severe anxiety.
Change in daytime sleepiness | 12 weeks
  Daytime sleepiness will be measured by a 8-item Epworth Sleepiness Scale (ESS). ESS is a widely used self-report questionnaire used to evaluate daytime sleepiness in the field of sleep medicine. Total score ranges from 0 to 24. Higher score indicates more daytime sleepiness.
Change in fatigue symptoms | 12 weeks
  Fatigue symptoms will be assessed by a 20-item Multidimensional Fatigue Inventory (MFI). MFI is a self-report questionnaire used to evaluate five dimensions of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Each dimension has four items. Total score of each dimension ranges from 4 to 20. Higher score indicates more severe fatigue for that dimension.
Change in sleep diary parameters | 12 weeks
  Consensus Sleep Diary (CSD) will be used to record sleep time, wake time and subjective sleeping quality daily. Parameters including sleep onset latency, time awake after sleep onset, total wake time, total sleep time and sleep efficiency will be calculated.
Change in gut microbiota composition | 12 weeks
  Relative abundance of gut bacteria at species level will be assessed by metagenomic analysis.
Change in gut microbiota diversity and richness | 12 weeks
  Species diversity (Shannon index) and richness (number of observed species) will be calculated based on the relative abundance of gut bacteria.
Similarity of gut microbiota composition to donor | 12 weeks
  Engraftment of donor species after intervention will be assessed by the similarity of gut microbiota composition to the donor.
Change in blood cytokine profile | 12 weeks
  Change in blood cytokine profile will be assessed, including levels of interferon gamma, interleukins, leptin, vascular endothelial growth factor, membrane-bound immunoglobulin, and tumour necrosis factor-α etc.
Change in blood cortisol | 12 weeks
  Change in blood cortisol will be assessed
Change in Melatonin level | 12 weeks
  Change in blood melatonin will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Whitaker M, Elliott J, Chadeau-Hyam M, Riley S, Darzi A, Cooke G, Ward H, Elliott P. Persistent COVID-19 symptoms in a community study of 606,434 people in England. Nat Commun. 2022 Apr 12;13(1):1957. doi: 10.1038/s41467-022-29521-z. PMID 35413949
- [Background] Tran VT, Porcher R, Pane I, Ravaud P. Course of post COVID-19 disease symptoms over time in the ComPaRe long COVID prospective e-cohort. Nat Commun. 2022 Apr 5;13(1):1812. doi: 10.1038/s41467-022-29513-z. PMID 35383197
- [Background] Liu Q, Mak JWY, Su Q, Yeoh YK, Lui GC, Ng SSS, Zhang F, Li AYL, Lu W, Hui DS, Chan PK, Chan FKL, Ng SC. Gut microbiota dynamics in a prospective cohort of patients with post-acute COVID-19 syndrome. Gut. 2022 Mar;71(3):544-552. doi: 10.1136/gutjnl-2021-325989. Epub 2022 Jan 26. PMID 35082169
- [Background] Li Y, Hao Y, Fan F, Zhang B. The Role of Microbiome in Insomnia, Circadian Disturbance and Depression. Front Psychiatry. 2018 Dec 5;9:669. doi: 10.3389/fpsyt.2018.00669. eCollection 2018. PMID 30568608
- [Background] Allegretti JR, Mullish BH, Kelly C, Fischer M. The evolution of the use of faecal microbiota transplantation and emerging therapeutic indications. Lancet. 2019 Aug 3;394(10196):420-431. doi: 10.1016/S0140-6736(19)31266-8. PMID 31379333
- [Background] Khoruts A, Sadowsky MJ. Understanding the mechanisms of faecal microbiota transplantation. Nat Rev Gastroenterol Hepatol. 2016 Sep;13(9):508-16. doi: 10.1038/nrgastro.2016.98. Epub 2016 Jun 22. PMID 27329806
- [Derived] Lau RI, Su Q, Ching JYL, Lui RN, Chan TT, Wong MTL, Lau LHS, Wing YK, Chan RNY, Kwok HYH, Ho AHY, Tse YK, Cheung CP, Li MKT, Siu WY, Liu C, Lu W, Wang Y, Chiu EOL, Cheong PK, Chan FKL, Ng SC. Fecal Microbiota Transplantation for Sleep Disturbance in Post-acute COVID-19 Syndrome. Clin Gastroenterol Hepatol. 2024 Dec;22(12):2487-2496.e6. doi: 10.1016/j.cgh.2024.06.004. Epub 2024 Jun 20. PMID 38908733